CLINICAL TRIAL: NCT01472731
Title: Guiding GC1008 Treatment of Primary Brain Tumors by 89Zr-GC1008 PET Imaging.
Brief Title: Safety and Imaging Study of GC1008 in Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC1008; 2010-021639-15 (EudraCT Number)
Record Dates: First submitted 2011-07-18; First posted 2011-11-16 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Primary Brain Tumors
Keywords: GC1008; PET imaging; primary brain tumors; recurrent high grade glioma's
MeSH Terms: conditions — Brain Neoplasms | interventions — fresolimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GC1008 imaging and treatment (Experimental): Part 1: Feasibility of 89Zr-GC1008 PET imaging in patients with suspicion of a malignant glioma to assess if GC1008 penetrates into the brain tumor and to quantify its uptake.
  Part 2: 89Zr-GC1008 PET imaging in patients with relapsed malignant glioma and phase II extension study with therapeutic GC1008 in these patients
  Interventions: Other: 89Zr-GC1008; Drug: GC1008

INTERVENTIONS:
Other: 89Zr-GC1008 — radioactive labeled GC1008, intravenous use, 37 MBq total
  Other Names: 89Zr-fresolimumab
Drug: GC1008 — 5 mg/kg intravenous use
  Other Names: fresolimumab

SUMMARY:
Brain tumors account for only 2% of all cancers but result in a disproportionate share of cancer morbidity and mortality. The five-year survival rates for the most common histologic subtypes, anaplastic astrocytoma and glioblastoma (glioblastoma multiforme, GBM), are 30% and 10%, respectively.

Drugs affecting transforming growth factor-β (TGF-β) might be of great interest for malignant glioma treatment. TGF-β is an oncogenic factor in advanced tumors where it induces proliferation, angiogenesis, invasion, and metastasis as well as suppresses the antitumoral immune response. In addition TGF-β and its TGF-β receptors, TβRI and TβRII, are overexpressed in GBMs. TGF-β signaling is involved in multiple steps of GBM development. GC1008 is an antibody that is capable of neutralizing TGF-β and may therefore offer a new treatment option for patients with malignant glioma.

For therapeutic success, it may be essential for GC1008 to reach the target site, in this case located in the brain. We will be able to prove this with 89Zr-GC1008 PET imaging. This imaging method also allows quantification of the amount of GC1008 reaching the tumor.

This study consists of 2 parts. In part 1, patients with a suspicion of a malignant glioma undergo an 89Zr-GC1008 PET scan before standard (surgical)treatment. In part 2, patients with relapsed malignant glioma will undergo an 89Zr-GC1008 PET scan and will be treated with GC1008 in a phase II study as there is no standard treatment for these patients.

We hypothesize that GC1008 uptake in brain tumors can be visualized and quantified using the 89Zr-GC1008 PET scan and GC1008 might offer a new treatment option for patients with relapsed malignant gliomas.

DETAILED DESCRIPTION:
Brain tumors account for only 2% of all cancers but result in a disproportionate share of cancer morbidity and mortality. The five-year survival rates for the most common histologic subtypes, anaplastic astrocytoma and glioblastoma (glioblastoma multiforme, GBM), are 30% and 10%, respectively.

After surgery, the standard treatment of malignant glioma is focused on cell death induction by DNA damage, neglecting the fact that invasion into surrounding brain tissue is a fundamental feature of and the major reason for treatment failure.

Drugs affecting transforming growth factor-β (TGF-β) might be of great interest for malignant glioma treatment. The reason for this is the fact that TGF-β acts as a tumor suppressor in normal epithelial cells and early-stage tumors but transforms in an oncogenic factor in advanced tumors where it induces proliferation, angiogenesis, invasion, and metastasis as well as suppresses the antitumoral immune response. In addition TGF-β expression and its TGF-β receptors, TβRI and TβRII, are overexpressed in GBMs. TGF-β signaling is involved in multiple steps of GBM development (Golestaneh, Mishra, 2005) and invasion (Wesolowska et al, 2008). Plasma TGF-β levels are elevated in GBM patients and decrease after surgical tumor resection (Schneider et al, 2006). Progression-free survival and overall survival are worse for malignant glioma patients with high TGF-β signaling compared with glioma patients with low TGF-β signaling activity (Bruna et al, 2007). All these features make TGF-β a promising target molecule for biological treatment approaches for GBM (Wick et al, 2006). Phase I/II-studies with the TGF-β2-specific antisense oligodeoxynucleotide AP12009 in malignant glioma showed promising results (Hau et al, 2007). Another approach to target TGF-β is with monoclonal antibodies, such as GC1008. GC1008 is a fully human IgG4 kappa monoclonal antibody capable of neutralizing all mammalian isoforms of TGF-β (i.e., 1, 2, and 3). For therapeutic success, it may be essential for GC1008 to reach the target site, in this case located in the brain. Our own data with 89Zr-bevacizumab, which is also an IgG, showed that the VEGF directed antibody bevacizumab penetrates the brain and is localized in brain metastases. We therefore expect GC1008 to reach the malignant glioma as well. In order to initiate clinical trials with TGF-β antibody in these patients it would clearly be of great help to prove that the drug arrives at the tumor site. 89Zr-GC1008 PET imaging will allow us to prove this. In addition, PET imaging allows quantification of the amount of GC1008 reaching the malignant glioma. A phase II study with GC1008 in patients with relapsed malignant gliomas will be initiated as currently, there is no standard treatment available for these patients.

Study objectives:

Part 1: Feasibility of 89Zr-GC1008 PET imaging in patients with suspicion of a malignant glioma to assess if GC1008 penetrates into the brain tumor and to quantify its uptake.

Part 2: 89Zr-GC1008 PET imaging in patients with relapsed malignant glioma and phase II extension study with therapeutic GC1008 in these patients.

For part 1, 12 patients will be included. For part 2, 12-20 patients will be included.

ELIGIBILITY:
Part 1

Inclusion Criteria

* > 18 years
* WHO 0,1,2
* Suspicion of malignant glioma on contrast-enhanced MRI
* Able to give written informed consent

Exclusion Criteria

* Meningeal carcinomatosis, uncontrolled seizures, or a disease that either causes or threatens neurologic compromise
* Pregnant or nursing women
* Known allergy to component of 89Zr-GC1008
* Significant medical or psychosocial problems

Part 2

Inclusion Criteria

* Relapsed malignant glioma
* Patient may have undergone surgery for the recurrence. Residual and measurable disease after surgery is not required. Surgery must have confirmed the recurrence. Post-operative MRI must be made within 48 hours following surgery
* For non operated patients, recurrent disease must be at least one bidimensionally measurable target lesion (contrast enhancing lesion) with one diameter of at least 2cm, based on MRI scan done within 4 weeks prior to start of treatment
* 18 years
* WHO 0,1,2
* Serum albumin ≥3.0 g/dL
* Adequate organ function including:

  * Hb ≥10.0 g/dL
  * ANC ≥1,500/mm3
  * platelets ≥100,000/mm3
  * Serum total bilirubin ≤1.5 x ULN (Patients with Gilbert's Disease may be included if their total bilirubin is ≤3.0 mg/dL)
  * ALT and AST ≤2.5 x ULN.
  * Estimated or measured creatinine clearance ≥60 mL/min
  * PT and PTT within normal ranges
* Negative tests for hepatitis viruses B and C and HIV, unless the result is consistent with prior vaccination or prior infection with full recovery
* Enrollment >4 weeks since major surgery, radiotherapy, chemotherapy (≥6 weeks if they were treated with a nitrosourea, mitomycin, or monoclonal antibodies), immunotherapy, or biotherapy/targeted therapies and recovered from the toxicity of prior treatment to ≤ Grade 1, exclusive of alopecia. Concurrent cancer therapy is not permitted (except for corticosteroids) (For long acting agents, a treatment free interval of 2 half lives should be considered)
* Able to give written informed consent
* Patients of child-producing potential must agree to use effective contraception while enrolled on study and receiving the experimental drug, and for at least 3 months after the last treatment

Exclusion Criteria

* History of ascites or pleural effusions , unless successfully treated, completely resolved, and the patient has not been treated for these conditions for >4 months
* Active thrombophlebitis, thromboembolism, hypercoagulability states, bleeding, or use of anti-coagulation therapy. Patients with a history of deep venous thrombosis may participate if successfully treated, completely resolved, and no treatment has been given for >4 months
* Hypercalcemia: Calcium >11.0 mg/dL (2.75 mmol/L) unresponsive or uncontrolled in response to standard therapy
* Pregnant or nursing women
* Diagnosis with another malignancy - unless following curative intent therapy, the patient has been disease free for at least 5 years and the probability of recurrence of the prior malignancy is <5%. Patients with curatively treated early stage squamous cell carcinoma of the skin, basal cell carcinoma of the skin, or cervical intraepithelial neoplasia are eligible for this study
* Organ transplant, including allogeneic bone marrow transplant
* Investigational agents used within 4 weeks prior to study enrollment (within 6 weeks for long-acting agents such as a monoclonal antibody)
* Immunosuppressive therapy including: cyclosporine A, tacrolimus, or sirolimus
* Significant or uncontrolled medical illness, such as congestive heart failure, myocardial infarction, symptomatic coronary artery disease, significant ventricular arrhythmias within the last 6 months, or significant pulmonary dysfunction. Patients with a remote history of asthma or active mild asthma may participate
* Active infection, including unexplained fever (temperature >38.1 'C), or antibiotic therapy within 1 week prior to enrollment
* Systemic autoimmune disease
* Known allergy to component of GC1008 or 89Zr-GC1008
* Significant medical or psychosocial problems

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-12; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Biomarker imaging | 2 years
  Part 1, Biomarker imaging: 89Zr-GC1008 PET imaging in patients with suspicion of a malignant glioma:
  Primary endpoint:
  - Quantification of uptake of 89Zr-GC1008 as determined by PET imaging. The data obtained from the PET-scans will be quantified as standardized uptake value (SUV).
Quantification of uptake | 2 years
  Part 2, In relapsed malignant glioma patients 89Zr-GC1008 PET imaging followed by participation in phase 2 study of GC1008
  Primary endpoint:
  - Quantification of uptake of 89Zr-GC1008 in relapsed malignant glioma patients as determined by PET imaging. The data obtained from the PET-scans will be quantified as standardized uptake value (SUV).

SECONDARY OUTCOMES:
Correlation of 89Zr-GC1008 tumor uptake | 2 years
  Part 1, Biomarker imaging: 89Zr-GC1008 PET imaging in patients with suspicion of a malignant glioma:
  Secondary endpoint:
  - Correlation of 89Zr-GC1008 tumor uptake with tumor histology, immunohistochemistry for TGF-β, VEGF expression, TGF-β tumor levels as determined by ELISA.
Correlation of 89Zr-GC1008 tumor uptake | 2 years
  Part 1, Biomarker imaging: 89Zr-GC1008 PET imaging in patients with suspicion of a malignant glioma:
  Secondary endpoint:
  - 89Zr-GC1008 biodistribution in humans.
Secondary endpoints Part 2 | 2 years
  * Radiological Response Rate; measured by conventional MRI
  * Overall survival (OS); assessed by clinical follow up
  * 6-month progression-free survival (PFS) rate; assessed by clinical follow up
  * Correlation of 89Zr-GC1008 tumor uptake pre-surgery and at relapse in the subgroup that underwent a 89Zr-GC1008 PET scan before primary surgery
  * Number of patients with a positive PET scan as determined by quantification of uptake of 89Zr-GC1008 in relapsed malignant glioma patients.
  * Correlation of 89Zr-GC1008 tumor uptake with treatment outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Annemiek ME Walenkamp, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands